CLINICAL TRIAL: NCT02690532
Title: The Role of Gut Permeability in Developing Celiac Disease and Non-Celiac Gluten Sensitivity
Brief Title: Gut Permeability Assessment in Celiac and Gluten Sensitive Children
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Imad Absah, M.D., Assistant Professor of Pediatrics, Mayo Clinic
Other Study IDs: 15-006018
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Celiac Disease
Keywords: Celiac; Gluten; Sensitivity; Permeability; Non-celiac gluten intolerance; Gastrointestinal Diseases; Digestive System Diseases
MeSH Terms: conditions — Celiac Disease; Hypersensitivity; Gastrointestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- High risk group: Children who are at high risk for developing celiac disease (siblings diagnosed with celiac disease).
- Non-celiac group: Children who are self-diagnosed with non-celiac gluten sensitivity.
- Control Group: Healthy control group (matched for age and gender).

SUMMARY:
This study will assess the effect of gluten on gut barrier function. Investigators at the Mayo Clinic have developed a new gut permeability test using rhamnose (sugar & water solution), and are hoping to prove its effectiveness in a clinical setting.

DETAILED DESCRIPTION:
The aim of this study is to assess effect of gluten on the gut barrier function in patients at high risk for celiac disease and non-celiac gluten sensitivity (NCGS) patients. This study will assess the gut permeability in three groups of patients 1) children who are at high risk for developing celiac disease (CD) (siblings of patients with celiac disease), 2) Children who are self-diagnosed with NCGS and 3) control group of patients matched for age and gender. Patients will undergo celiac serologic and genetic testing, after which the rhamnose test will be performed to assess the presence of increased gut permeability.

ELIGIBILITY:
High Risk group:

* Sibling with a confirmed diagnosis of celiac disease
* No history Celiac disease or any other bowel disease

Non-Celiac Gluten Sensitivity group:

* Self-diagnosis of gluten sensitivity
* No history of celiac disease or other bowel disease

Healthy group:

* Absence of celiac disease or any other bowel disease
* No sensitivity to gluten

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of three groups of children, aged 2-17 years. The first group will be children with siblings that have celiac disease, the second group will be children with non-celiac gluten sensitivity and the third group will be healthy children.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Gut Permeability | Baseline
  Assess the effect of gluten on gut permeability in children at high risk of developing celiac disease or gluten sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Imad Absah, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No